CLINICAL TRIAL: NCT00902408
Title: The Effect of Lutein-enriched-egg Beverage on Progression of Age-related Macular Degeneration, a Randomized Trial
Brief Title: Effect of Lutein-enriched-egg Beverage on Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Newtricious (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MEC 07-1-127
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lutein (Experimental): Lutein enriched eggs
  Interventions: Dietary Supplement: Lutein enriched eggs
- Placebo (Placebo Comparator): Non enriched
  Interventions: Dietary Supplement: Lutein enriched eggs

INTERVENTIONS:
Dietary Supplement: Lutein enriched eggs — 1 year of daily enriched lutein eggs or placebo

SUMMARY:
After a pilot trial where we showed an substantial increase in plasma lutein levels and a increase in macular pigment optical density after only 3 months of daily consumption of a lutein-enriched egg-beverage, we now propose to study the effect these changes have on subjects with early ( undiagnosed) stages of macular degeneration. Age-related macula degeneration, is the leading cause of blindness in many developed countries[1-6] in older persons (usually over 55 years of age). Visual compromise rises exponentially after age of 70[7] with a 5-year incidence of around 1%. The incidence of bilateral AMD in persons with unilateral late ARM observed over a period of 10 years of over 50% with a 2.1-2.8% overall incidence in study population[8]. To date there is no curative way of fighting AMD. With the results of this trial we hope to show that with daily consumption of these enriched beverage, we can slow the progression of AMD. (Protocol page 8-10)

DETAILED DESCRIPTION:
Rationale: In our pilot study (MEC 07-1-127) we saw an increase in both plasma as macular levels of lutein and zeaxanthin. Current believe is that this increase might help against the further deterioration of the retina seen in age-related macular degeneration (AMD) by scavenging for free radicals and filtering out harmful blue light rays[1, 2]. For the purpose of establishing whether these believes hold some truth, we want now to investigate the effect of lutein and zeaxanthin increase in subject with early signs of AMD on visual acuity, visual field and contrast sensibility. To relate these results to our previous study we will also measure the changes in plasma and macular concentrations of these xanthophylls. Once more we will be using the egg-beverage from the pilot study. These have been proven safe and showed no changes in lipid levels after 3 months of consumption.

Objective: To assess whether there is the same increase in macular pigment optical density as in healthy subject and to see if there is any change in visual function after a year of intervention.

Study design: This will be a randomized, double blind, placebo controlled, interventional trial. Subjects will be randomized, stratified for gender and age, into two groups (N=50 each) receiving either the intervention product (base on 1.5 yolk of a lutein enriched egg containing 0.921 ± 0.106mg of lutein and 0.137 ± 0.014mg of zeaxanthin per yolk) or a placebo. Subject will be followed for 1 year and will be seen three times for measurements.

Study population: 100 subjects, ages 50 and older with drusen and/or Retinal pigment epithelium (RPE) alterations on retinal image.

Main study parameters/endpoints: Changes in amount of early macular degeneration signs on fundus photographs. Macular pigment optical density. Plasma lutein and zeaxanthin levels.

Nature and extend of the burden and risks associated with participation, benefit and group relatedness: Subjects will be seen three times with a total of 22 ( + 1 hour screening) hours. Methods used in this trial are commonly used techniques which have been proven safe in either previous trials or clinical practice. Subjects' sight will be limited for the investigated eye for a few hours after every visit because of the use of Tropicamide, this is standard practice at our ophthalmology department with only sporadic, and treatable side effects (acute angle-closure glaucoma in 0.03%). Subjects in the intervention group are expected to show a slower progression of the disease than those in the placebo group. We will be using the same egg-beverage as in the pilot study which showed no changes in lipid levels.

ELIGIBILITY:
Inclusion Criteria:

* Early signs of AMD on fundus photographs (drusen and or retinal pigment epithelium alterations in at least one eye)
* 50 years and older
* Vision > 0.5
* Non-smoker
* No ocular media opacity
* Uses no nutritional supplements containing Lutein or Zeaxanthin
* BMI < 30
* No known cardiovascular disease

Exclusion Criteria:

* Diabetes
* Known lipid metabolism disease
* Blood lipid level modifiers (e.g. Statin)
* Known allergy to eggs or egg products

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in amount of early macular degeneration signs on fundus photographs. Macular pigment optical density. Plasma lutein and zeaxanthin levels. | 1 year

SECONDARY OUTCOMES:
Assessing morphological changes of the retina, visual acuity, contrast sensitivity, field of vision, and rod function. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elton Kellly, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Eye Clinic Maastrich, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] van der Made SM, Kelly ER, Berendschot TT, Kijlstra A, Lutjohann D, Plat J. Consuming a buttermilk drink containing lutein-enriched egg yolk daily for 1 year increased plasma lutein but did not affect serum lipid or lipoprotein concentrations in adults with early signs of age-related macular degeneration. J Nutr. 2014 Sep;144(9):1370-7. doi: 10.3945/jn.114.195503. Epub 2014 Jul 2. PMID 24991045